CLINICAL TRIAL: NCT03161535
Title: Effectiveness of a Rehabilitation Program in Improving Sleep Quality, Emotional Distress, Circadian Rhythms, and Quality of Life in Patients With Esophageal Cancer
Brief Title: Effectiveness of a Rehabilitation Program in Improving Quality of Life in Patients With Esophageal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-04-001A
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Exercise; Nutrition Assessment; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): The rehabilitation program was composed of two parts: an exercise program and a diet-teaching program. The exercise program was a 12-week home-based program that comprised moderate-intensity brisk walking for 40 min per session, with 3 sessions per week; in addition, weekly exercise counseling was provided through telephone. The diet teaching program was provided to the patients by using a diet booklet at baseline (same timing as the exercise program), and its contents were used to instruct the patients regarding dietary principles to be followed.
  Interventions: Other: exercise and dietary education; Other: weekly telephone consultations concerning exercise and diet.
- usual-care group (No Intervention): The control group (CG) received usual care, whereas a nurse, the manager for esophageal cancer treatment, provided routine care, conducted follow-ups, and offered information on esophageal cancer to the experimental group (EG).

INTERVENTIONS:
Other: exercise and dietary education — 1. A 12-week regimen of home-based walking exercises, comprising walking at a moderate intensity for 40 min, three times a week, was administered along with weekly exercise counseling. After collecting pretrial measurements, we explained the participants how to perform the exercises, according to an instruction manual for the exercise regimen. The detailed instructions, provided at the hospital clinics, included the determination of activity intensity, demonstration of pulse measurement, criteria for scores of 6-20 on the Borg's rating of perceived exertion (RPE), prevention of exercise-related injuries, and conditions necessitating termination of an exercise session. Participants were instructed that the exercises would be effective only if they reached 60%-80% of the target heart rate, as determined by the Karvonen method, and 13-15 on the RPE.
  2. Diet-teaching program (using dietary education booklet).
  Arms: exercise group
Other: weekly telephone consultations concerning exercise and diet. — For each participant, we discussed exercise regimen-related issues and diet weekly through the telephone. For instance, we discussed whether participants' exercise fulfilled the prescribed intensity, duration, or frequency and whether the participants experienced any adverse effects.
  Arms: exercise group

SUMMARY:
This study will investigate the effectiveness of a rehabilitation program in improving sleep quality, emotional distress, circadian rhythms, and quality of life in patients with esophageal cancer in Taiwan.

Hypothesis:

1. The quality of life in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, 24th, and 36th month.
2. The quality of sleep in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, 24th, and 36th month.
3. The emotional distress in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, 24th, and 36th month.
4. The circadian rhythms in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, 24th, and 36th month.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of a rehabilitation program in improving sleep quality, emotional distress, circadian rhythms, and quality of life in patients with esophageal cancer in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophageal cancer who were aged ≥20 years, could communicate in either Mandarin or Taiwanese, and were not cognitively impaired were included.

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Quality of life (EORTC QLQ-C30 ) | baseline
  using European Organization for Research and Treatment cancer QLQ-C30 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-C30 ) | 3rd month after recruited
  using European Organization for Research and Treatment cancer QLQ-C30 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-C30 ) | 6th month after recruited
  using European Organization for Research and Treatment cancer QLQ-C30 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-C30 ) | 12th month after recruited
  using European Organization for Research and Treatment cancer QLQ-C30 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-C30 ) | 24th month after recruited
  using European Organization for Research and Treatment cancer QLQ-C30 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-C30 ) | 36th month after recruited
  using European Organization for Research and Treatment cancer QLQ-C30 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-OES 18 ) | baseline
  using European Organization for Research and Treatment cancer QLQ-OES 18 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-OES 18 ) | 3rd month after recruited
  using European Organization for Research and Treatment cancer QLQ-OES 18 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-OES 18 ) | 6th month after recruited
  using European Organization for Research and Treatment cancer QLQ-OES 18 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-OES 18 ) | 12th month after recruited
  using European Organization for Research and Treatment cancer QLQ-OES 18 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-OES 18 ) | 24th month after recruited
  using European Organization for Research and Treatment cancer QLQ-OES 18 (EORTC) to measure quality of life.
Quality of life (EORTC QLQ-OES 18 ) | 36th month after recruited
  using European Organization for Research and Treatment cancer QLQ-OES 18 (EORTC) to measure quality of life.

SECONDARY OUTCOMES:
Subjective sleep quality | baseline
  using Pittsburgh Sleep Quality Index
Subjective sleep quality | 3rd month after recruited
  using Pittsburgh Sleep Quality Index
Subjective sleep quality | 6th month after recruited
  using Pittsburgh Sleep Quality Index
Subjective sleep quality | 12th month after recruited
  using Pittsburgh Sleep Quality Index
Subjective sleep quality | 24th month after recruited
  using Pittsburgh Sleep Quality Index
Subjective sleep quality | 36th month after recruited
  using Pittsburgh Sleep Quality Index
Objective sleep quality | baseline
  using Actigraph for measure Objective sleep quality
Objective sleep quality | 3rd month after recruited
  using Actigraph for measure Objective sleep quality
Objective sleep quality | 6th month after recruited
  using Actigraph for measure Objective sleep quality
Objective sleep quality | 12th month after recruited
  using Actigraph for measure Objective sleep quality
Objective sleep quality | 24th month after recruited
  using Actigraph for measure Objective sleep quality
Objective sleep quality | 36th month after recruited
  using Actigraph for measure Objective sleep quality
Emotional distress | baseline, 3rd month, 6th month, 12th month, 24th month, and 36th month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Circadian rhythms | baseline, 3rd month, 6th month, 12th month, 24th month, and 36th month after recruited
  Circadian rhythms including 24-h autocorrelation coefficient (r24) and in bed less than out of bed dichotomy index (I<O) collection from actigraphy.

OTHER OUTCOMES:
Recurrence status | Third month (T2), sixth month (T3), twelfth month (T4), twenty-fourth month (T5), and thirty-sixth month (T6).
  Recurrence status was assessed through chart review.
Nutritional status | Baseline (T1), third month (T2), sixth month (T3), twelfth month (T4), twenty-fourth month (T5), and thirty-sixth month (T6)
  Nutritional status, including body weight, Body Mass Index (BMI), and serum albumin level, was assessed through chart review. However, patients will not be required to return to the hospital for blood tests; only existing blood test reports available in the medical records will be retrieved.
Survival status | Third month (T2), sixth month (T3), twelfth month (T4), twenty-fourth month (T5), and thirty-sixth month (T6).
  Survival status was assessed through chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences; YU-CHUNG WU, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

REFERENCES:
- [Derived] Chen HM, Huang CS, Wu YC, Chien LI, Hsu PK. The effects of a 3-month walking and dietary education program on the quality of life of patients with esophageal cancer: a 1-year follow-up randomized controlled trial. Support Care Cancer. 2025 May 1;33(5):441. doi: 10.1007/s00520-025-09489-4. PMID 40312569
- [Derived] Chen HM, Lin YY, Wu YC, Huang CS, Hsu PK, Chien LI, Lin YJ, Huang HL. Effects of Rehabilitation Program on Quality of Life, Sleep, Rest-Activity Rhythms, Anxiety, and Depression of Patients With Esophageal Cancer: A Pilot Randomized Controlled Trial. Cancer Nurs. 2022 Mar-Apr 01;45(2):E582-E593. doi: 10.1097/NCC.0000000000000953. PMID 33813524